CLINICAL TRIAL: NCT06734884
Title: Efficacy and Safety of Anti-interleukin 5 Receptor Therapy (Benralizumab) in Patients With Drug Reaction With Eosinophilia and Systemic Symptoms (DRESS)
Brief Title: Interest of a Targeted Therapy for the Treatment of a Severe Form of Hypersensitivity to Drug (DRESS Syndrome)
Acronym: BENRADRESS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020_57; 2022-502750-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-23; First posted 2024-12-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: DRESS Syndrome
Keywords: DRESS syndrome; drug hypersensitivity; Eosinophil; Benralizumab; targeted therapy
MeSH Terms: conditions — Drug Hypersensitivity Syndrome; Drug Hypersensitivity | interventions — benralizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benralizumab (Experimental)
  Interventions: Drug: Benralizumab 30 MG/ML [Fasenra]
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator: Placebo-Control Arm 0.9% Sodium Chloride

INTERVENTIONS:
Drug: Benralizumab 30 MG/ML [Fasenra] — Subcutaneous injection 30 mg at day 2, week 4 and week 8.
  Arms: Benralizumab
Drug: Placebo Comparator: Placebo-Control Arm 0.9% Sodium Chloride — Subcutaneous injection at day 2, week 4 and week 8
  Arms: Placebo

SUMMARY:
Drug Reaction with eosinophilia and Systemic Symptoms (DRESS) is a rare and severe multiorgan drug reaction whose pathophysiological mechanisms underlying remain unclear, but may involve the role of several immune cells like eosinophils. iIndeed,the number of eosinophils is increased in blood and/or in organs tiisues in at least 50% of patients with DRESS. There is no specific treatment available. The standard of care is corticosteroids, but they may be inefficient or poorly tolerated. The aim of this research is to find out whether a specific treatment of the immunological response in DRESS syndrome would be useful in combination with corticosteroids to speed up the recovery from DRESS syndrome and therefore reduce the total length of your hospital stay when your illness is being managed. This a multicenter, international, prospective, interventional study, double-blinded, placebo-controlled, randomized, in two balanced parallel groups, one receiving the standard of care (topical or systemic corticosteroids, according to the severity of DRESS syndrome) and the other one corticsoteroids and a targeted therapy against eosinophils (benralizumab, already available in other eosinophilic diseases like asthma).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (minimum 18year-old)
2. diagnosed at D0 (= baseline and inclusion) with DRESS defined by:

   1. with a REGIScar score at D0 calculated at at least 4 (4 or 5: probable DRESS; >5: definite case of DRESS), see Annex: REGIScar criteria
   2. Skin eruption with an onset considered as compatible with a DRESS syndrome according to the investigator's opinion after the uptake of one or several drug(s)
   3. AND Fever ≥ 38°C at the time of the examination or notion of a thermal peak ≥ 38°C in the preceding 72 hours.
   4. At least 1 organ disorder compatible with the diagnosis of DRESS syndrome among the following disorders:

      * Adenopathies present in at least 2 different sites and ≥ 1 cm in size
      * Acute hepatitis defined by :

        * Elevation of liver enzymes in serum: ALAT (Alanine Aminotransferase) and/or ASAT (Aspartate Aminotransferase)
        * AND/OR an increase in serum total bilirubin, according to the standards of the local analysis laboratory (in the absence of a history of liver disease: ASAT and/or ALAT ≥ 3N (=3 times normal)
        * AND/OR total bilirubin ≥ 2N
      * Acute renal failure defined by :

        * An increase in creatinine according to local laboratory standards
        * AND a sterile cytobacteriological examination (in the absence of a history of renal disease: creatininaemia ≥ 1.5N
        * AND/OR increase in creatinine ≥ 0.3 mg/dl (or ≥ 26.5 mol/L)
        * AND/OR urine output < 0.3 ml/kg/h (over ≥ 24h).
      * Pulmonary impairment defined by:

        * Oxygen saturation (SpO2) measured by pulse oximetry ≤ 95% in room air
        * And/or the presence of an interstitial syndrome on a standard chest X-ray or a CT scan of the chest (in the absence of any other cause of lung damage).
3. With eosinophilia (blood eosinophil count ≥ 500/mm3 or ≥0.5 G/L).
4. Patient having given written informed consent
5. patient with social insurance

Exclusion Criteria:

1. Patients <18 year-old
2. Patients with DRESS with REGIScar score <4
3. Patients without skin eruption at baseline
4. Eosinophils blood count <500/mm3 or < 0.5 G/L at baseline
5. Patients with contra-indication to blood samples dedicated to the biocollection, according to the investigator's opinion
6. Patients with contra-indication to stop the culprit drug(s) involved in DRESS
7. Past history of hypersensitivity to biological drugs
8. Patients who received a previous anti-IL5 or anti-IL5 receptor therapy within 5 half lives (= 4 months) before inclusion
9. Patients with a contra-indication of topical corticosteroids (mainly a past history of contact eczema with clobetasol propionate)
10. Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2029-01-05 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Efficacity of an add-on treatment with benralizumab to decrease the total hospitalization for DRESS duration within a 52 weeks (W52) period in patients diagnosed with DRESS syndrome and treated with corticosteroids (CS) | from inclusion to 52 weeks
  Number of days spent in hospital for the management of DRESS syndrome

SECONDARY OUTCOMES:
Percentage of body surface with cutaneous lesions due to DRESS and severity grade of skin involvement observed within the 52 weeks period | at Day4, Day 7, Week 2, Week 4, Week 12, Week 24 and Week 52
  Percentage of body surface with cutaneous lesions recorded
Number and severity grade of organ lesions due to DRESS observed within the 52 weeks period | Total number of organ lesions within 52 weeks. These organ lesions will be recorded at Day 4, Day7, Week 2, Week 4, Week 12, Week 24 and Week 52.
Dosage of blood eosinophils during the 52 weeks after inclusion | number of cells per mm3 or per liter) performed at baseline (D0 = prior treatment), and at Day 2, Day 4, Day 7, Week 2, Week 4, Week 8, Week 12, Week 24, Week 52.
Number of flares or relapses of DRESS during a 52 week-period after inclusion | Total number of exacerbation/worsening or occurrence/reappearance of DRESS signs identified within the Week 52 period and recorded at Day 2, Day 4, Day 7, Week 2, Week 4, Week 8, Week 12, Week 24, Week 52.
Consumption of topical or systemic corticosteroids during a 52 week-period after inclusion | Total quantity of superpotent topical or systemic corticosteroids (CS) used at Day 7, Week 2, Week 4, Week 8, Week 12, Week 24, Week 52
  expressed in weight in grammes

CONTACTS AND LOCATIONS:
Locations (1):
- Delphine STAUMONT-SALLE, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF